CLINICAL TRIAL: NCT06439771
Title: A Multicenter, Open-Label, Phase 2 Study to Evaluate the Efficacy, Safety and Pharmacokinetics of YL202 in Patients With Locally Advanced or Metastatic Breast Cancer With TNBC, HR-Positive, HER2-Zero-expression or HER2-Low-expression
Brief Title: A Phase 2 Study to Evaluate the Efficacy, Safety and Pharmacokinetics of YL202 in Patients With BC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MediLink Therapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YL202-CN-202-01
Record Dates: First submitted 2024-05-16; First posted 2024-06-03 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-06

CONDITIONS: Locally Advanced or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Experimental: Corhort A (Experimental): YL202 is provided as the lyophilized powder, 200 mg/vial. Triple-negative breast cancer (TNBC) patients will be given YL202 by intravenously once every 3 weeks (Q3W) as a cycle.
  Interventions: Drug: YL202 should be intravenously infused
- Experimental: Corhort B (Experimental): YL202 is provided as the lyophilized powder, 200 mg/vial. HR-positive breast cancer with HER2-Zero-expression and HER2-Low-expression patients will be given YL202 by intravenously once every 3 weeks (Q3W) as a cycle.
  Interventions: Drug: YL202 should be intravenously infused
- Experimental: Corhort C (Experimental): YL202 is provided as the lyophilized powder, 200 mg/vial. Breast cancer patients who have previously failed treatments of HER2-ADC or TROP2-ADC (excluding HER2+ patients, ie, HER2 IHC 3+ or IHC 2+/ISH+ patients) will be given YL202 by intravenously once every 3 weeks (Q3W) as a cycle.
  Interventions: Drug: YL202 should be intravenously infused

INTERVENTIONS:
Drug: YL202 should be intravenously infused — For each patient, YL202 should be intravenously infused over 60±10 min.

SUMMARY:
This study is a multicenter, open-label, phase 2 clinical study to evaluate the efficacy, safety and pharmacokinetics of YL202 in patients with locally advanced or metastatic breast cancer with TNBC, HR-positive, HER2-zero-expression or HER2-low-expression

ELIGIBILITY:
Inclusion Criteria:

1. Have been informed of the study before the start of the study and voluntarily sign name and date on the informed consent form.
2. Patients with locally advanced or metastatic disease (according to the UICC and AJCC staging system [Version 8]) who are not candidates for curative surgery or radiotherapy.
3. Patients who are pathologically confirmed advanced/unresectable or metastatic breast cancer with HR-negative and HER2-negative,.
4. Patients who are confirmed HR positive and HER2-Zero-expression and HER2-Low-expression.
5. Breast cancer patients who have previously failed treatments of HER2-ADC or TROP2-ADC.
6. Have at least 1 extracranial measurable lesion as a target lesion per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
7. Have Adequate organ and bone marrow function within 7 days prior to the first dose.
8. Female patients of childbearing potential must agree to use highly effective contraception from screening throughout the duration of the study and for at least 6 months after the last dose of study drug.
9. Have a expected survival ≥ 3 months.
10. Have ability and willingness to comply with protocol-specified visits and procedures.

Exclusion Criteria:

1. Have prior treatment with an agent targeting HER3.
2. Have prior intolerance to treatment with topoisomerase I inhibitor or an ADC that consists of topoisomerase I inhibitor.
3. Have been enrolled in another clinical study concurrently unless it is an observational clinical study or in the follow-up phase of an interventional study.
4. Have insufficient washout period for prior anticancer therapy prior to first dose of the study drug.
5. Have major surgery (excluding diagnostic surgery) within 4 weeks prior to the first dose of study drug or anticipation of major surgery during the study.
6. Have prior allogeneic bone marrow transplant or prior solid organ transplant.
7. Have received treatment with systemic steroids.
8. Have received any live vaccine within 4 weeks prior to the first dose of study drug or intend to receive a live vaccine during the study.
9. Leptomeningeal metastases or carcinomatous meningitis, spinal cord compression.
10. Brain metastases with the exceptions.
11. Have uncontrolled or clinically significant cardiovascular and cerebrovascular disease.
12. Have clinically significant concomitant pulmonary diseases.
13. Have a diagnosis of Gilbert's syndrome.
14. Have pleural effusion, abdominal effusion.
15. Have a history of gastrointestinal perforation and or fistula within 6 months prior to the first dose.
16. Have serious infection.
17. Patients with human immunodeficiency virus (HIV) infection.
18. Have active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
19. Have any other primary malignancy within 5 years prior to the first dose of study drug.
20. Have unresolved toxicities from prior anticancer therapy.
21. Have a history of severe hypersensitivity reactions to the drug substance, inactive ingredients in the drug product, or other monoclonal antibodies.
22. Lactating women, or women who are confirmed to be pregnant by pregnancy test within 3 days prior to the first dose.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2028-07-29 (Estimated)

PRIMARY OUTCOMES:
ORR assessed according to RECIST v1.1 | By the end of trial date, approximately within 36 months
  ORR: defined as the proportion of patients who achieved a best overall response of complete response (CR) or partial response (PR).
Determination of the recommended dose of YL202 in the pivotal clinical study | By the end of trial date, approximately within 36 months

SECONDARY OUTCOMES:
Progression-free survival (PFS) assessed according to RECIST v1.1 | By the end of trial date, approximately within 36 months
Clinical benefit rate (CBR) assessed based on RECIST v1.1 | By the end of trial date, approximately within 36 months
Depth of response (DpR) assessed based on RECIST v1.1 | By the end of trial date, approximately within 36 months
Disease control rate (DCR) assessed based on RECIST v1.1 | By the end of trial date, approximately within 36 months
Duration of response (DOR) assessed based on RECIST v1.1 | By the end of trial date, approximately within 36 months
Time to response (TTR) assessed based on RECIST v1.1 | By the end of trial date, approximately within 36 months
Evaluate the overall survival (OS) | By the end of trial date, approximately within 36 months
Adverse event (AE), described in terms of type, frequency, severity, time, and relationship with study treatment | Approximately within 36 months
Characterize the PK parameter AUC | Approximately within 36 months
  steady-state area under curve (AUC)
Characterize the PK parameter Cmax | Approximately within 36 months
  peak concentration (Cmax)
Characterize the PK parameter Ctrough | Approximately within 36 months
  trough concentration (Ctrough)
Characterize the PK parameter CL | Approximately within 36 months
  clearance (CL)
Characterize the PK parameter Vd | Approximately within 36 months
  volume of distribution (Vd)
Characterize the PK parameter t1/2 | Approximately within 36 months
  half-life (t1/2)
Incidence of anti-YL202 antibody | Approximately within 36 months
Evaluate the corelaton between different levels of HER3 expression and the sum of CR rate, PR rate and SD rate | Approximately within 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China